CLINICAL TRIAL: NCT06329401
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2b Study Evaluating the Safety and Efficacy of Pirfenidone Solution for Inhalation (AP01) in Participants With PPF
Brief Title: A Study Evaluating the Safety and Efficacy of Inhaled AP01 in Participants With Progressive Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Avalyn Pharma Inc. (Industry)
Collaborators: DevPro Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP01-007
Record Dates: First submitted 2024-03-12; First posted 2024-03-25 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Progressive Pulmonary Fibrosis
Keywords: Chronic-Fibrosing-ILD with progressive phenotype, PF-ILD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AP01 High Dose BID (Experimental): Pirfenidone Solution for Inhalation
  Interventions: Drug: AP01
- AP01 Low Dose BID (Experimental): Pirfenidone Solution for Inhalation
  Interventions: Drug: AP01
- Placebo BID (Placebo Comparator): Placebo solution for inhalation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AP01 — Oral inhalation solution
  Other Names: Pirfenidone Solution
  Arms: AP01 High Dose BID; AP01 Low Dose BID
Other: Placebo — Placebo oral inhalation solution
  Arms: Placebo BID

SUMMARY:
A randomized, double-blind, placebo-controlled clinical study to evaluate the safety and efficacy of 2 doses of inhaled pirfenidone (AP01) versus placebo on top of standard of care in participants with PPF over 52 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled clinical study to evaluate the safety and efficacy of 2 doses of AP01 (pirfenidone solution for inhalation) versus placebo on top of standard of care in participants with PPF over 52 weeks. Up to 300 eligible participants will be randomized to 1 of 3 treatment arms: AP01 high dose, AP01 low dose, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participant meets criteria for PPF, as follows:
* In subjects with interstitial lung disease (ILD) of known or unknown etiology other than idiopathic pulmonary fibrosis (IPF) who have radiological evidence of pulmonary fibrosis, PPF is defined as:

Physiological evidence of disease progression with at least 1 of the following criteria despite treatment with approved or unapproved medications commonly used in practice (per Investigator):

1. Relative decline in FVC ≥10% predicted within the previous 24 months based on documented historical spirometry assessments
2. Relative decline in FVC ≥5% to <10% predicted within the previous 24 months based on documented historical spirometry assessments with at least 1 of the 2 following criteria:

   * Worsening respiratory symptoms (Note: Changes attributable to comorbidities e.g., infection, heart failure must be excluded) OR
   * Radiological (HRCT) evidence of disease progression per a local or central radiologist (from historical HRCT taken up to 24 months prior to Screening Visit 1), for example:

     * Increased extent or severity of traction bronchiectasis and bronchiolectasis
     * New ground-glass opacity with traction bronchiectasis
     * New fine reticulation
     * Increased extent or increased coarseness of reticular abnormality
     * New or increased honeycombing
     * Increased lobar volume loss
3. Worsening of respiratory symptoms (Note: Changes attributable to comorbidities e.g., infection, heart failure must be excluded) AND radiological (HRCT) evidence of disease progression per a local or central radiologist

   * Meeting all of the following criteria during the Screening Period:

a. FVC ≥45% of predicted normal at Screening Visit 1, b. Forced expiratory volume at 1 second (FEV1)/FVC ≥0.7 or ≥age-adjusted lower limit of normal at Screening Visit 1, c. Diffusing capacity of lung for carbon monoxide (DLCO) ≥30% of predicted, corrected for hemoglobin at Screening Visit 1, d. Acceptability: Participants can perform acceptable spirometry (i.e., meet American Thoracic Society (ATS)/ European Respiratory Society (ERS) acceptability criteria at both Screening Visits).

• For subjects already on nintedanib (up to 30% of subjects): Must have been on nintedanib for at least 6 months prior to Screening with or without dose adjustments and/or drug interruptions during that period. For subjects who have discontinued nintedanib prior to Screening: Must have been off of nintedanib for a minimum of 12 weeks.

Exclusion Criteria:

* Current treatment with oral pirfenidone or treatment with oral pirfenidone within 3 months prior to Screening.
* Elevated liver enzymes and liver injury at Screening defined as:

  1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ˃ 3 times the upper limit of normal (ULN)
  2. Bilirubin >2.0 x ULN
* Renal disease with a creatinine clearance < 30 mL/min, calculated according to the Chronic Kidney Disease Epidemiology Collaboration formula. Retesting is allowed once.
* Diagnosis of idiopathic pulmonary fibrosis (IPF) based on the ATS diagnostic algorithm for IPF. UIP that is not idiopathic, for example related to rheumatoid arthritis (RA), familial interstitial lung disease (ILD), or other is not exclusionary.
* Greater extent of emphysema than of fibrotic ILD on HRCT. Note: CT results must be confirmed through the central over read process.
* Significant clinical worsening of PPF between Screening
* Participants who cannot meet protocol-specified Baseline stability criteria. FVC Baseline stability is defined as the FVC assessments at Visit 3 being within ±12% of the mean of the FVC assessments obtained at the 2 preceding visits. At Visit 3, if the pre-dose FVC is outside of ±12% range, the participant will not be randomized and will be considered a screen failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of AP01 high dose twice a day (BID) or AP01 low dose twice a day (BID) compared to placebo twice a day (BID) | Week 52
  Change from baseline in forced vital capacity (FVC) (mL)

SECONDARY OUTCOMES:
To evaluate the effect of AP01 high dose and AP01 low dose compared to placebo on disease progression (defined as absolute FVC percent predicted decline of ≥10% prior to Week 52) | 52 weeks
  Time to disease progression
To evaluate the effect of AP01 high dose, AP01 low dose compared to placebo on quality of life (QoL) | 52 weeks
  Absolute change from Baseline in QoL measurements as assessed by Living with Pulmonary Fibrosis Symptoms and Impact Questionnaire (L-PF) total score. The L-PF is a 44-item questionnaire to assess how impacted a participant is by disease symptoms on a scale from 0 (Not at all) to 4 (Extremely). The higher the summary score, the greater the impairment.
To evaluate the change from baseline in quantitative lung fibrosis score. | 52 weeks
  Change in lung fibrosis score.

OTHER OUTCOMES:
To evaluate the safety of AP01 high dose and AP01 low dose compared to placebo | 52 weeks
  Incidents of adverse events (AEs), serious adverse events (SAEs), and treatment-emergent deaths

CONTACTS AND LOCATIONS:
Overall Officials: Avalyn Pharma, Inc., Study Director — Avalyn Pharma Inc.
Locations (146):
- United States (60):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pulmonary Associates, PA, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai, Los Angeles, California
  - UCLA, Los Angeles, California
  - Newport Native MD, Inc., Newport Beach, California
  - Paradigm Clinical Research - Redding, Redding, California
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - UCONN Health, Farmington, Connecticut
  - Yale University, New Haven, Connecticut
  - Clinical Site Partners, LCC, Leesburg, Florida
  - Renstar Medical Research, Ocala, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - SEC Clinical Research, Pensacola, Florida
  - Clinical Site Partners, Winter Park, Florida
  - Piedmont Healthcare, Inc., Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Endeavor Health, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Hannibal Regional Healthcare System, Hannibal, Missouri
  - Northwell Health - Mount Kisco, Mount Kisco, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Pulmonix, Greensboro, North Carolina
  - Piedmont HealthCare, PA, Statesville, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Summit Health, Bend, Oregon
  - The Oregon Clinic Pulmonary East, Portland, Oregon
  - The Oregon Clinic Pulmonary West, Portland, Oregon
  - The Pennsylvania State University, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Vanderbilt Lung Institute, Nashville, Tennessee
  - Baylor Scott & White Research Institute, Baylor University Medical Center, Dallas, Texas
  - El Paso Pulmonary Association, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center, Houston, Texas
  - Metroplex Pulmonary and Sleep Center, PA, McKinney, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - Inova Healthcare, Falls Church, Virginia
  - University of Washington, Seattle, Washington
- Argentina (8):
  - Fundacion Respirar, Buenos Aires, Buenos Aires
  - CINME, Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Ave Pulmo, Fundacion Enfisema, Mar del Plata, Buenos Aires
  - Centro Respiratorio Quilmes, Quilmes, Buenos Aires
  - Instituto de Medicina Respiratoria, Córdoba, Córdoba Province
  - CIMER Centro Integral de Medicina Respiratoria, San Miguel de Tucumán, Tucumán Province
  - Investigaciones En Patologias Respiratorias, San Miguel de Tucumán, Tucumán Province
- Australia (10):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Lung & Sleep, Kingswood, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Macquarie University Clinical Trials Unit, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Institute for Respiratory Health, Nedlands, Perth West Australia
  - Wallace Street Specialist Centre/Lung Research QLD Pty Ltd, Brisbane, Queensland
  - Lung Research Victoria, Footscray, Victoria
  - Alfred Health, Melbourne, Victoria
  - Canberra Hospital, Canberra
- Canada (6):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Dynamic Drug Advancement, Ajax, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Research Institute McGill University Health Center, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec-Université Laval, Québec, Quebec
  - CIC Mauricie, Trois-Rivières, Quebec
- France (9):
  - CHU de Rennes, Rennes, Cedex NA
  - CHU Tours, Tours, Indre et Loire
  - Robert Schuman Hospital UNEOS, Metz, Lorraine
  - Louis Pradel Hospital, Lyon, Lyon
  - University of Montpellier, Montpellier, Montpellier
  - CHU Angers, Angers
  - APHP - Hopital Bicetre, Le Kremlin-Bicêtre
  - Hôpital Paris St Jozeph, Paris
  - Hôpital Haut-Lévêque, Pessac
- Germany (8):
  - Pneumologisches Studienzentrum München-West, Munich, Bavaria
  - RoMed Klinikum Rosenheim, Rosenheim, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Studienzentrum Dr. Claus Keller, Frankfurt, Main Hessia
  - Ruhrlandklinik Essen, Klinik fuer Pneumologie, Essen, North Rhine-Westphalia
  - Universitätsmedizin Mainz - Zentrum für Thoraxerkrankungen, Mainz, Rhineland-Palatinate
  - Uniklinikum Leipzig Medizinische Klinik II - Bereich, Leipzig, Saxony
  - Vivantes Klinikum Neukölln - Klinik für Innere Medizin - Pneumologie und Infektiologie, Berlin, State of Berlin
- Italy (9):
  - A.O.U. delle Marche - Ospedale di Torrette, Torrette, Ancona
  - Azienda Ospedaliera dei Colli - Ospedale Monaldi, Naples, Campania
  - Università degli Studi di Napoli Federico II - Ospedale Monaldi, Napoli, Campania
  - IRCCS AOU di Bologna - Policlinico Sant' Orsola, Bologna, Emilia-Romagna
  - Azienda Sanitaria Universitaria Giuliano Isontina, Venezia, Giulia
  - Fondazione IRCCS Policlinico San Matteo - UOC Pneumologia, Pavia, Lombardy
  - Ospedale San Giuseppe, Milan, Milano
  - HUMANITAS Research Hospital, Rozzano, Milano
  - A.O.U. Policlinico G. Rodolico, Catania, Sicily
- Erasmus University Medical Center, Rotterdam, Netherlands
- New Zealand (4):
  - Greenlane Clinical Centre, Auckland, Auckland
  - Health New Zealand, Christchurch, Canterbury
  - Dunedin Hospital, Dunedin, Dunedine
  - Bay of Plenty Clinical School, Tauranga, South Tauranga
- Poland (4):
  - Vitamed Galaj I Cichomski sp.j., Bydgoszcz, Bydgoszc
  - University Hospital in Krakow, Krakow, Krakow
  - PRYWATNY GABINET LEKARSKI GINEKOLOGIA I POŁOZNICTWO ULTRASONOGRAFIA Prof. Dr hab. Med. Jacek Suzin, Lodz
  - AppleTreeClinics Network, Lodz, Łódź Voivodeship
- Spain (10):
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital de Sant Pau y la Santa Creu, Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Universitary de Bellvitge, Barcelona
  - Hospital Universitario Puerta del Mar - Leon-Jimenez, Cadiz
- Turkey (Türkiye) (3):
  - Ege University Medical Faculty Hospital, Bornova, İzmir
  - Cukurova University Medical Faculty, Adana
  - Health Sciences University, Gulhane Faculty of Medicine, Ankara
- United Kingdom (14):
  - Hull University Teaching Hospital NHS Trust, Cottingham, East Yorkshire
  - Birmingham Heartlands Hospital, Birmingham, Heartlands
  - Leicester Biomedical Research Centre - Respiratory Theme, Glenfield, Leicester
  - St George's University Hospitals NHS Foundation Trust, London, London
  - ILD Unit, University Hospitals Birmingham NHS Foundation Trust Theme, Birmingham, Midlands
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxon
  - Royal Devon, Exeter, South West
  - The Royal Wolverhampton NHS Trust, New Cross Hospital, Research and Development, Wolverhampton, West Midlands
  - St James University Hospital - LTHT, Leeds, West Yorkshire
  - Royal Papworth Hospital, Cambridge
  - Royal Brompton Hospital, London
  - Manchester University NHS Foundation Trust, Manchester
  - Nottingham University NHS Trust, Nottingham
  - University Hospitals of North Midlands NHS Trust, Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] West A, Chaudhuri N, Barczyk A, Wilsher ML, Hopkins P, Glaspole I, Corte TJ, Sterclova M, Veale A, Jassem E, Wijsenbeek MS, Grainge C, Piotrowski W, Raghu G, Shaffer ML, Nair D, Freeman L, Otto K, Montgomery AB. Inhaled pirfenidone solution (AP01) for IPF: a randomised, open-label, dose-response trial. Thorax. 2023 Sep;78(9):882-889. doi: 10.1136/thorax-2022-219391. Epub 2023 Mar 22. PMID 36948586
- [Derived] Kolb M, Corte TJ, Feldman J, Nathan SD, Reisner C, Nair D, Woodhead F, Lazarus H, Conoscenti C. Design of the MIST study: a double-blind, randomised, placebo-controlled phase 2b trial of pirfenidone solution for inhalation in patients with progressive pulmonary fibrosis. BMJ Open Respir Res. 2025 Dec 25;12(1):e003059. doi: 10.1136/bmjresp-2024-003059. PMID 41448793
- See also: Content — http://thorax.bmj.com/content/78/9/882.long